CLINICAL TRIAL: NCT02553694
Title: Impact of a Short Educational Video on OSA Patient Satisfaction, Knowledge and Outcomes
Brief Title: Sleep Apnea Video Education for CPAP (SAVE-CPAP)
Acronym: SAVE-CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB14-0198
Record Dates: First submitted 2014-08-05; First posted 2015-09-17 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA, Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Enhanced education and Enhanced follow up (Experimental): Subjects will watch a short video and will be contacted by an MD by phone
  Interventions: Other: Enhanced education; Other: Usual follow up
- Usual education and Usual follow up (Active Comparator): Standard education by American Academy of Sleep Medicine (AASM)- created educational pamphlets and will be contacted by a sleep center staff member by phone
  Interventions: Other: Usual education; Other: Enhanced follow up
- Enhanced education and Usual follow up (Experimental): Subjects will watch a short video immediately prior to the initiation of the in-laboratory polysomnogram and will be contacted by sleep center non-MD staff member by phone
  Interventions: Other: Enhanced education; Other: Enhanced follow up
- Usual education with Enhanced follow up (Experimental): Standard education by American Academy of Sleep Medicine (AASM)- created educational pamphlets and contacted by an MD by phone
  Interventions: Other: Usual education; Other: Usual follow up

INTERVENTIONS:
Other: Enhanced education — Investigator created video to help educate subject before the in-laboratory split night polysomnogram. The subject will watch the short video immediately prior to the initiation of the in-laboratory polysomnogram.
  Arms: Enhanced education and Enhanced follow up; Enhanced education and Usual follow up
Other: Usual education — Usual education by American Academy of Sleep Medicine (AASM)- created educational pamphlets
  Arms: Usual education and Usual follow up; Usual education with Enhanced follow up
Other: Usual follow up — MD will follow up by phone after the in-laboratory split night polysomnogram
  Arms: Enhanced education and Enhanced follow up; Usual education with Enhanced follow up
Other: Enhanced follow up — Sleep center non-MD staff member will follow up by phone after the in-laboratory split night polysomnogram
  Arms: Enhanced education and Usual follow up; Usual education and Usual follow up

SUMMARY:
The purpose of this study is to determine how satisfied patients are when undergoing an overnight polysomnogram (sleep study), what their knowledge about sleep apnea is, and what factors affect obstructive sleep apnea (OSA) treatment use.

DETAILED DESCRIPTION:
The effects of educational interventions on subject compliance, satisfaction, and knowledge of their condition will be examined through the use of video vs pamphlet and MD vs staff contact for follow-up visit reminder.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years of age who are referred to the University of Chicago sleep laboratory for split-night polysomnography by a non-sleep physician and who have a consultation appointment with a sleep physician following the appointment
* Have not had prior contact with a sleep physician or prior exposure to CPAP therapy.

Exclusion Criteria: Subjects will be excluded for any of the following characteristics: -Non-English speaking

* Illiterate
* Sleep study is negative for sleep apnea (apnea-hypopnea index < 5 events/hr)
* Subject does not undergo CPAP titration during the in-laboratory polysomnogram
* Subject does not have a working telephone number
* Poor eyesight or hearing
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
CPAP Therapy Adherence | 30 days post in-lab split night polysomnogram
  Subject use of CPAP device will be monitored electronically. Subjects will be randomized to educational intervention of either viewing a video or reading a pamphlet prior to in-laboratory split night polysomnogram (sleep study) and initiation of CPAP therapy, and CPAP adherence rates of the two groups will be compared and reported.

SECONDARY OUTCOMES:
Subject compliance with sleep clinic appointment | within 3 months after the in-laboratory split night polysomnogram
  Subjects will be randomized to receive a reminder call for follow up clinic appointment either from MD or staff, and the compliance rates of the two groups will be compared based on call type and educational intervention type.
Patient Knowledge About Sleep Apnea and CPAP Therapy | 1 day post in-laboratory split night polysomnogram
  Subjects will be administered 2 questionnaires which measure knowledge about their condition, both before and after the in-laboratory split night polysomnogram (sleep study). The scores of the two questionnaires will be combined for both test administrations. Subjects will be randomized to educational intervention of either viewing a video or reading a pamphlet prior to sleep study and initiation of CPAP therapy, and the change in the combined questionnaire scores of the two groups will be compared and reported.
Patient Satisfaction With the in-laboratory split night polysomnogram | 1 day post in-laboratory split night polysomnogram
  Subjects will be administered 2 questionnaires which measure their mood and well-being, both before and after the in-laboratory split night polysomnogram. The questionnaires will be scored and the scores for each subject will be combined at both testing administrations. On the night of the in-laboratory polysomnogram subjects will be randomized to educational intervention of either viewing a video or reading a pamphlet prior to the initiation of the polysomnogram and initiation of CPAP therapy, and the change in the combined questionnaire scores of the two groups will be compared and reported.
CPAP Therapy Adherence | 1 month post sleep clinic visit or the date of the missed sleep clinic visit
  Subjects will be randomized to receive a reminder call for follow up sleep clinic appointment either from MD or non-MD sleep center staff, and the compliance rates of the two groups will be compared based on call type and educational intervention type.

CONTACTS AND LOCATIONS:
Overall Officials: Babak Mokhlesi, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohli P, Balachandran JS, Malhotra A. Obstructive sleep apnea and the risk for cardiovascular disease. Curr Atheroscler Rep. 2011 Apr;13(2):138-46. doi: 10.1007/s11883-011-0161-8. PMID 21253882
- [Background] Metabolic disorders associated with obstructive sleep apnea in adults. Adv Cardiol. 2011;46:67-138. doi: 10.1159/000325106. Epub 2011 Oct 13. PMID 22005190
- [Background] Balachandran JS, Yu X, Wroblewski K, Mokhlesi B. A brief survey of patients' first impression after CPAP titration predicts future CPAP adherence: a pilot study. J Clin Sleep Med. 2013 Mar 15;9(3):199-205. doi: 10.5664/jcsm.2476. PMID 23493772
- [Derived] Guralnick AS, Balachandran JS, Szutenbach S, Adley K, Emami L, Mohammadi M, Farnan JM, Arora VM, Mokhlesi B. Educational video to improve CPAP use in patients with obstructive sleep apnoea at risk for poor adherence: a randomised controlled trial. Thorax. 2017 Dec;72(12):1132-1139. doi: 10.1136/thoraxjnl-2017-210106. Epub 2017 Jun 30. PMID 28667231